CLINICAL TRIAL: NCT04921943
Title: Hypertonic Saline for Treatment of Pulmonary Mycobacterium Avium Complex (MAC) Disease
Brief Title: Hypertonic Saline for MAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: NTM Info & Research, Inc. (Unknown); University Health Network, Toronto (Other); New York University (Other)
Responsible Party: Principal Investigator, Kevin Winthrop, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAC-HS
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Nontuberculous Mycobacterial Lung Disease; Nontuberculous Mycobacterium Infection
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — Saline Solution, Hypertonic; Azithromycin; Ethambutol; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hypertonic saline (Experimental): Patients who randomize to the hypertonic saline arm will be prescribed a nebulizer device to nebulize hypertonic saline (7%) twice daily for 12 weeks. Hypertonic saline (3%) can be prescribed in the case of poor tolerability of the 7% solution.
  Interventions: Drug: Hypertonic saline
- Standard of Care (Active Comparator): Patients who randomize to the standard of care arm will receive treatment for pulmonary MAC based on the approved ATS/IDSA guidelines. Changes to standard of care regimen may be made based on the investigator's discretion.
  Interventions: Drug: Azithromycin; Drug: Ethambutol; Drug: Rifampin

INTERVENTIONS:
Drug: Hypertonic saline — Nebulizing with 7% hypertonic saline twice daily for 12 weeks.
  Arms: Hypertonic saline
Drug: Azithromycin — Standard of care
  Arms: Standard of Care
Drug: Ethambutol — Standard of care
  Arms: Standard of Care
Drug: Rifampin — Standard of care
  Arms: Standard of Care

SUMMARY:
The MAC-HS study is a testing whether hypertonic saline helps improve symptoms and clearance of mycobacteria in patients with M. avium complex lung infections.

DETAILED DESCRIPTION:
The MAC-HS study is an open label, randomized control trial of hypertonic saline in pulmonary M. avium complex patients. Eligible patients who consent to participate will be randomized 1:1 to hypertonic saline or standard of care for 12 weeks. All patients in the treatment group will take inhaled hypertonic saline twice daily for 12 weeks. Patients may continue with other airway clearance methods (i.e. flutter, acapella valve, aerobika, postural drainage, huff cough, percussion). Patients may also be treated with antibiotics targeted at other pathogens if an exacerbation occurs. Patients may also be actively treated with inhaled corticosteroid at the time of enrollment, with dosing adjustments during the trial discouraged. Patients with disease progression at any time can be discontinued from the study treatment and treated according to ATS/IDSA guidelines at the discretion of the primary investigator. However, such patients will still complete the 12 week final visit, sputum collection and AE assessment.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 positive MAC sputum cultures in the last 12 months with at least one AFB positive sputum obtained within 12 weeks prior to randomization
* Meet American Thoracic Society (ATS)/ Infectious Disease Society of America (IDSA) 2007 pulmonary clinical disease criteria[1]
* Age 18 and older
* Diagnosis of Bronchiectasis and/or bronchiectatic findings evident on chest CT report
* Ability to provide informed consent

Exclusion Criteria:

* Any patient who is unwilling or unable to provide consent or to comply with this protocol
* Cavitary NTM disease
* Patients who are currently taking or within the prior 6 months received any of the following: bedaquiline, or any component of ATS/IDSA multi-drug recommended therapy (macrolide, ethambutol, rifampin) for MAC treatment
* Diagnosis of HIV
* Diagnosis of Cystic fibrosis
* Active pulmonary tuberculosis, fungal, or nocardial disease requiring treatment at screening
* Current use of chronic systemic corticosteroids at doses of 15 mg/day for more than 3 months
* Prior lung or other solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Culture conversion | 12 weeks
  At least two negative AFB cultures on different days.

SECONDARY OUTCOMES:
Semi-quantitative culture results | 12 weeks
  Evaluate acid fast bacilli (AFB) smear results to see if there is a decreased mycobacterial load (i.e. AFB smear 4+ decreasing to 3+).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - NYU Langone Health, New York, New York
  - Oregon Health & Science University, Portland, Oregon
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No